CLINICAL TRIAL: NCT02413008
Title: A Phase II Prospective, Randomized, Double-Blind, Placebo-Controlled and Multi-Centre Clinical Trial to Assess the Safety of 0.005 % Estriol Vaginal Gel in Hormone Receptor-Positive Postmenopausal Women With Early Stage Breast Cancer in Treatment With Aromatase Inhibitor in the Adjuvant Setting
Brief Title: A Clinical Trial to Assess the Safety of 0.005 % Estriol Vaginal Gel in Hormone Receptor-Positive Postmenopausal Women With Early Stage Breast Cancer in Treatment With Aromatase Inhibitor in the Adjuvant Setting
Acronym: BLISSAFE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ITF Research Pharma, S.L.U. (Industry)
Collaborators: Spanish Breast Cancer Research Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITFE-2026-C10; 2014-004517-84 (EudraCT Number)
Record Dates: First submitted 2015-04-01; First posted 2015-04-09 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-06

CONDITIONS: Vaginal Atrophy
Keywords: vaginal atrophy; breast cancer; vaginal dryness; aromatase inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — Estriol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.005% estriol vaginal gel (Experimental): Route: Vaginal. Administration by an applicator inserted deep inside the vagina Dose: 1 g of gel, containing 50 Mcg of estriol Dosage schedule: Weeks 1-3: single daily application Weeks 4-12: twice weekly administration
  Interventions: Drug: estriol
- placebo vaginal gel (Placebo Comparator): Route: Vaginal. Administration by an applicator inserted deep inside the vagina Dose: 1 g of gel. Dosage schedule: Weeks 1-3: single daily application Weeks 4-12: twice weekly administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: estriol — 0.005% estriol vaginal gel
  Other Names: Blissel (estriol); Gelistrol (estriol)
  Arms: 0.005% estriol vaginal gel
Drug: Placebo — placebo vaginal gel
  Arms: placebo vaginal gel

SUMMARY:
This is a phase II, prospective, randomized, double-blind, placebo-controlled, international (Spain and Sweden) and multicentre study to explore the safety of 0.005% estriol vaginal gel in women with early stage breast cancer in treatment with Non-Steroidal Aromatase Inhibitors (NSAIs) in the adjuvant setting and symptoms of vaginal atrophy.

DETAILED DESCRIPTION:
This is a phase II, prospective, randomized, double-blind, placebo-controlled, international (Spain and Sweden) and multicentre study.

In the setting of postmenopausal hormone receptor positive breast cancer, treatment with aromatase inhibitors (AIs) is the most effective and well-studied therapy. Vaginal dryness is one of the most frequently reported symptom caused by this adjuvant therapy which may lead to a reduced adherence in breast cancer women.

This study will explore the safety of 0.005% estriol vaginal gel in this oncological context, to demonstrate that this medicinal product is a safe option to treat the vaginal atrophy caused by AIs, without a clinically relevant influence in gonadotropins or systemic estrogen levels.

The main objective is to evaluate the levels of Follicle Stimulating Hormone (FSH) after treatment with 0.005% estriol vaginal gel in hormone receptor-positive postmenopausal women with early stage breast cancer in treatment with Non-Steroidal Aromatase Inhibitors (NSAIs) in the adjuvant setting and symptoms of vaginal atrophy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to beginning specific protocol procedures.
2. Patients must have histological confirmation of breast adenocarcinoma with stage I-IIIA, documented at a local pathology department.
3. The breast tumors must be estrogen-receptor positive and/or progesterone receptor positive (≥1% of stained tumor cells by Immunohistochemistry (IHC) as determined by the local laboratory) with any Human Epidermal Growth Factor Receptor 2(HER2) status.
4. Postmenopausal status defined as: 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 Milli-international units per milliliter (mIU/ml) or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
5. Patient must be receiving the non-steroidal aromatase inhibitors anastrozole or letrozole as breast cancer treatment in the adjuvant setting for a minimum of 6 months.
6. Women suffering from moderate to severe vaginal dryness according to the FDA guidelines for drug development in postmenopausal women (Center for Drug Evaluation and Research, (CDER) Jan 2003). A moderate symptom will be considered if the symptom is present, bothersome and annoying, and a severe symptom will be considered if the symptom is present, bothersome and annoying, and interferes with the normal patient activity.
7. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
8. Adequate bone marrow as defined by the following laboratory values:

   1. Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L.
   2. Platelets (plt) ≥ 100 x 109/L.
   3. Hemoglobin (Hgb) ≥ 10 g/dl.
9. Patient has adequate organ function as defined by the following laboratory values:

   1. Serum creatinine ≤ 1.5 x Upper Limit of Normal (ULN).
   2. Bilirubin ≤ 1.5 × ULN.
   3. Alkaline phosphatase ≤ 2 × ULN.
   4. Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2 × ULN.
10. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. Stage IIIB-IV breast cancer or bilateral breast cancer.
2. Treatment with any other current anti-tumoral therapy (chemotherapy, anti-Her2…etc) besides the NSAI. Pamidronate or Alendronate are permitted.
3. Prior history of other malignancy within 5 years of study entry, aside from non-melanoma skin cancer or carcinoma-in-situ of the uterine cervix adequately treated.
4. Postmenopausal uterine bleeding. Vaginal bleeding of unknown etiology.
5. Patients with endometrial thickness equal to or greater than 4 mm measured by transvaginal ultrasound.
6. Patients who have received any type of vulvovaginal treatment in the 15 days prior to the start of the study.
7. Use of any hormone, natural (phytoestrogens) or herbal products for the treatment of menopausal symptoms within the last 3 months.
8. Current or previous history of thromboembolic disease or coagulopathies.
9. Severe cardiovascular or respiratory diseases in the previous 6 months.
10. Renal Impairment.
11. Hepatitis B and/or hepatitis C carriers (unless with normal hepatic function).
12. Known human immunodeficiency virus infection.
13. Known hypersensitivity to NSAI.
14. Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
15. Previous investigational treatment for any condition or participation in any clinical trial within 4 weeks of inclusion date.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-10-16 (Actual); Primary Completion 2017-02-10 (Actual); Study Completion 2017-02-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., L'Hospitalet de Llobregat, Barcelona
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., A Coruña
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., Jaén
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., Madrid
  - For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., Valencia
- For additional information regarding investigative sites for this trial, contact ITF Research Pharma S.L.U., Stockholm, Sweden

REFERENCES:
- [Derived] Sanchez-Rovira P, Hirschberg AL, Gil-Gil M, Bermejo-De Las Heras B, Nieto-Magro C. A Phase II Prospective, Randomized, Double-Blind, Placebo-Controlled and Multicenter Clinical Trial to Assess the Safety of 0.005% Estriol Vaginal Gel in Hormone Receptor-Positive Postmenopausal Women with Early Stage Breast Cancer in Treatment with Aromatase Inhibitor in the Adjuvant Setting. Oncologist. 2020 Dec;25(12):e1846-1854. doi: 10.1634/theoncologist.2020-0417. Epub 2020 Jun 9. PMID 32459035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study had an initial safety phase of the trial started on March 30th, 2015; the treatment phase of the trial started in October 16th, 2015 and the study ended globally on February 10th, 2017
Pre-assignment Details: After Inform Consent signature and prior randomization the following data was collected for subject's eligibility: Medical and surgical history and demographics; physical examination, ECOG PS, hematology, blood chemistry, urine test, transvaginal ultrasound, Blood (serum) samples for FSH and LH determination and evaluation of vaginal dryness.
Groups:
- Placebo Vaginal Gel: Route: Vaginal. Administration by an applicator inserted deep inside the vagina Dose: 1 g of gel. Dosage schedule: Weeks 1-3: single daily application Weeks 4-12: twice weekly administration
  Placebo
Period: Overall Study
Arm/Group | 0.005% Estriol Vaginal Gel | Placebo Vaginal Gel
Started | 50 | 11
Completed | 43 | 9
Not Completed | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- 0.005% Estriol Vaginal Gel: Route: Vaginal. Administration by an applicator inserted deep inside the vagina Dose: 1 g of gel, containing 50 Mcg of estriol Dosage schedule: Weeks 1-3: single daily application Weeks 4-12: twice weekly administration
  estriol
- Total: Total of all reporting groups
Arm/Group | 0.005% Estriol Vaginal Gel | Placebo Vaginal Gel | Total
Number analyzed (Participants) | 50 | 11 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 9 | 55
  >=65 years | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (7.6) | 61.4 (4.7) | 59.3 (7.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 50 | 11 | 61
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 17 | 4 | 21
  Spain | 33 | 7 | 40

OUTCOME MEASURES:

1. Primary Outcome: Variation in Serum Levels of Follicle Stimulating Hormone (FSH)
Description: Change from Baseline (mean screening-baseline) to Week 12 in Serum Levels of Follicle Stimulating Hormone (FSH) compare to natural physiological variability (screening-baseline variation)
Time Frame: from baseline to 12 weeks of treatment
Population: postmenopausal participants
Measure: Median (Inter-Quartile Range); unit: mIU/ml
Arm/Group | 0.005% Estriol Vaginal Gel | Placebo Vaginal Gel
Number analyzed (Participants) | 50 | 11
mIU/ml | -2.8 [-13.1 to 7.4] | 1.4 [-5.4 to 15.7]
Statistical Analysis 1: Comparison: 0.005% Estriol Vaginal Gel; The variations of the levels of FSH after treatment was studied in each women at baseline, week 3 and week12 weeks, the variation of levels between two arms were analysed using a non-parametric test Mann-Whitney-Wilcoxon. The intra individual variation (differences between the pre study determinations screening and baseline) was compared to the variation between baseline and the values obtained at every study visit; Test type: Other — The primary endpoint, the variation of FSH between week 12 and baseline and also comparing by arm will be analyzed using a non-parametric test (Mann-Whitney-Wilcoxon test); p = 0.10, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo Vaginal Gel; The variations in the intensities for each one of the symptoms and signs of the vaginal atrophy, after 3 and 12 weeks, in each treatment arm, will be compared using the non-parametric test Mann-Whitney-Wilcoxon; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.413, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Test type: Other; p = 0.15, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Variation in Serum Levels of FSH at Week 1, Week 3 and Week 8
Description: Change from Baseline (mean screening-baseline) to Week 1, Week 3 and Week 8 in Serum Levels of Follicle Stimulating Hormone (FSH) compare to natural physiological variability ( screening-baseline variation)
Time Frame: Change from baseline to week 1, week 3 and week 8
Population: postmenopausal women
Measure: Mean (Inter-Quartile Range); unit: mIU/ml
Arm/Group | 0.005% Estriol Vaginal Gel | Placebo Vaginal Gel
Number analyzed (Participants) | 50 | 11
mIU/ml
  change from baseline to week 1 | -4.8 [-11.6 to 2.6] | 4.2 [-7.8 to 7.3]
  change from baseline to week 3 | -4.2 [-12.0 to 3.5] | -0.9 [-4.0 to 2.3]
  change from baseline to week 8 | -2.6 [-10.1 to 7.9] | 5.2 [-11.8 to 9]
Statistical Analysis 1: Comparison: 0.005% Estriol Vaginal Gel; Variation in serum levels of FSH at week 1; Test type: Other; p < 0.05, Dunn Test
Statistical Analysis 2: Comparison: 0.005% Estriol Vaginal Gel; Variation in serum levels of FSH at week 3; Test type: Other; p < 0.05, Dunn Test
Statistical Analysis 3: Comparison: 0.005% Estriol Vaginal Gel; Variation in serum levels of FSH at week 8; Test type: Other; p > 0.05, Dunn Test

3. Secondary Outcome: Variation in Serum Levels of Luteinizing Hormone (LH)
Description: Change from (mean screening-baseline) in plasma levels of LH to Week 1, Week 3, Week 8 and Week 12 in Serum Levels of LH compare to natural physiological variability ( screening-baseline variation)
Time Frame: Change from baseline to week 1, week 3, week 8 and week 12
Population: postmenopausal women
Measure: Median (Inter-Quartile Range); unit: mIU/ml
Arm/Group | 0.005% Estriol Vaginal Gel | Placebo Vaginal Gel
Number analyzed (Participants) | 50 | 11
mIU/ml
  change from LH baseline to week 1 | -0.6 [-3.7 to 2.8] | 0.2 [-1.8 to 8.1]
  change from LH baseline to week 3 | -0.5 [-4.1 to 3.5] | 0.3 [-1.8 to 7.7]
  change from LH baseline to week 8 | -0.3 [-4.9 to 3.1] | -1.3 [-2.0 to 6.0]
  change from LH baseline to week 12 | -0.8 [-5.3 to 2.9] | 1.3 [-1.6 to 7.1]
Statistical Analysis 1: Comparison: 0.005% Estriol Vaginal Gel; Change in serum levels of Luteinizing hormone (LH) from baseline to week 1; Test type: Other; p > 0.05, Dunn Test
Statistical Analysis 2: Comparison: 0.005% Estriol Vaginal Gel; Change in serum levels of Luteinizing hormone (LH) from baseline to week 3; Test type: Other; p > 0.05, Dunn Test
Statistical Analysis 3: Comparison: 0.005% Estriol Vaginal Gel; Change in serum levels of Luteinizing hormone (LH) from baseline to week 8; Test type: Other; p > 0.05, Dunn Test
Statistical Analysis 4: Comparison: 0.005% Estriol Vaginal Gel; Change in serum levels of Luteinizing hormone (LH) from baseline to week 12; Test type: Other; p = 0.135, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Variation in Plasma Levels of Estriol
Description: Change in plasma levels of estriol at weeks 1, 3, 8 and 12 compared to baseline
Time Frame: Change from baseline to week 1, week 3, week 8 and week 12
Population: postmenopausal women
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | 0.005% Estriol Vaginal Gel | Placebo Vaginal Gel
Number analyzed (Participants) | 50 | 11
pg/mL
  Change between baseline and week 1 | -1.7 [-10.7 to 0.0] | 0.0 [0.0 to 0.0]
  Change between baseline and week 3 | 0.0 [-3.4 to 0.5] | 0.0 [0.0 to 0.0]
  Change between baseline and week 8 | 0.0 [-5.0 to 0.5] | 0.0 [0.0 to 0.0]
  Change between baseline and week 12 | 0.0 [-6.8 to 0.5] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Change from baseline to week 1 in plasma levels of estriol; Test type: Other; p = 0.043, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Change from baseline to week 3 in plasma levels of estriol; Test type: Other; p = 0.649, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Change from baseline to week 8 in plasma levels of estriol; Test type: Other; p = 0.588, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Change from baseline to week 12 in plasma levels of estriol; Test type: Other; p = 0.67, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Variation in Plasma Levels of Estradiol
Description: Change in plasma levels of estradiol at weeks 1, 3, 8 and 12 compared to baseline.
Time Frame: Change from baseline to week 1, week 3, week 8 and week 12
Population: postmenopausal women
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | 0.005% Estriol Vaginal Gel | Placebo Vaginal Gel
Number analyzed (Participants) | 50 | 11
pg/mL
  Change between baseline and week 1 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Change between baseline and week 3 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Change between baseline and week 8 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Change between baseline and week 12 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Change from baseline to week 1 in plasma levels of estradiol; Test type: Other; p = 0.342, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Change from baseline to week 3 in plasma levels of estradiol; Test type: Other; p = 0.523, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Change in plasma levels of estradiol from baseline to week 8; Test type: Other; p = 0.523, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Change in plasma levels of estradiol from baseline to week 12; Test type: Other; p = 0.163, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Variation in Plasma Levels of Estrona
Description: Change in plasma levels of estrona at weeks 1, 3, 8 and 12 compared to baseline.
Time Frame: Change from baseline to week 1, week 3, week 8 and week 12
Population: postmenopausal women
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | 0.005% Estriol Vaginal Gel | Placebo Vaginal Gel
Number analyzed (Participants) | 50 | 11
pg/mL
  Change from baseline to week 1 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Change between baseline and week 3 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  change from baseline to week 8 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Change from baseline to week 12 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Change in plasma levels of estrona from baseline to week 1; Test type: Other; p = 0.418, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Change in plasma levels of estrona from baseline to week 3; Test type: Other; p = 0.642, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Change in plasma levels of estrona from baseline to week 8; Test type: Other; p = 0.175, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Change in plasma levels of estrona from baseline to week 12; Test type: Other; p = 0.084, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Changes in Vaginal pH Between Baseline and Week 3 and Week 12
Description: Measurement of vaginal pH on the vaginal secretion using a reactive strip and compare pH value between baseline and the diferent timepoints
Time Frame: week 3 and week 12 vs baseline
Population: postmenopausal women
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | 0.005% Estriol Vaginal Gel | Placebo Vaginal Gel
Number analyzed (Participants) | 50 | 11
units on a scale
  Change from baseline to Week 3 | 2.0 [0.5 to 2.5] | 0.5 [-0.5 to 1.0]
  Change from baseline to Week 12 | 1.3 [0.5 to 2.5] | 0.5 [0.0 to 1.5]
Statistical Analysis 1: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Change in pH between baseline and week 3; Test type: Other; p < 0.01, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Change in pH between baseline and week 12; Test type: Other; p = 0.057, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Changes in Dyspareunia
Description: Changes in dyspareunia from baseline to week 3 and week 12 Each symptom will be scored in a numeric scale from 0 to 3, as shown 0 Absence. The symptom is not present
  1. The symptom is of mild intensity, without interfering in the patient's activity
  2. The symptom is of moderate intensity, causing obvious discomfort to the patient
  3. The symptom is stated as very irritating and severe in intensity
Time Frame: week 3 and week 12 vs baseline
Population: postmenopausal women
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 0.005% Estriol Vaginal Gel | Placebo Vaginal Gel
Number analyzed (Participants) | 50 | 11
score on a scale
  Change between baseline and week 3 | 1.0 [1.0 to 2.0] | 1.0 [0.0 to 1.0]
  Change between baseline and week 12 | 2.0 [1.0 to 2.5] | 1.0 [0.0 to 2.0]
Statistical Analysis 1: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Changes in dyspareunia from baseline to week 3; Test type: Other; p = 0.14, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Changes in dyspareunia from baseline to week 12; Test type: Other; p = 0.25, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change in Pruritus or Itching From Baseline to Week 3 and Week 12
Description: Change in pruritus or itching from baseline to week 3 and week 12
  Each symptom will be scored in a numeric scale from 0 to 3, as shown below:
  0 Absence. The symptom is not present
  1. The symptom is of mild intensity, without interfering in the patient's activity
  2. The symptom is of moderate intensity, causing obvious discomfort to the patient
  3. The symptom is stated as very irritating and severe in intensity
Time Frame: Change from baseline to week 3 and week 12
Population: postmenopausal women
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | 0.005% Estriol Vaginal Gel | Placebo Vaginal Gel
Number analyzed (Participants) | 50 | 11
units on a scale
  Changes between baseline and week 3 | 0.0 [0.0 to 1.0] | 0.0 [-1.0 to 2.0]
  Changes between baseline and week 12 | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 1.0]
Statistical Analysis 1: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Change from baseline to week 3; Test type: Other; p = 0.28, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Change from baseline to week 12; Test type: Other; p = 0.34, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Changes in Vaginal Dryness
Description: Change in vaginal dryness puntuation score from baseline to w3 and w12
  Each symptom will be scored in a numeric scale from 0 to 3, as shown below:
  0 Absence. The symptom is not present
  1. The symptom is of mild intensity, without interfering in the patient's activity
  2. The symptom is of moderate intensity, causing obvious discomfort to the patient
  3. The symptom is stated as very irritating and severe in intensity
Time Frame: week 3 and week 12 vs baseline
Population: postmenopausal women
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | 0.005% Estriol Vaginal Gel | Placebo Vaginal Gel
Number analyzed (Participants) | 50 | 11
units on a scale
  Change between baseline and week 3 | 1.0 [1.0 to 2.0] | 1.0 [0.0 to 1.0]
  Change between baseline and week 12 | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0]
Statistical Analysis 1: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Changes in vaginal dryness from baseline to week 3; Test type: Other; p = 0.14, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Changes in vaginal dryness from baseline to week 12; Test type: Other; p < 0.01, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Changes in Total Score of Symptoms of Vaginal Atrophy
Description: Changes in Symptoms of vaginal atrophy (vaginal dryness, dyspareunia and pruritus) at week 3 and week 12 vs baseline.
  Each symptom will be scored in a numeric scale from 0 to 3, as shown below:
  0 Absence. The symptom is not present
  1. The symptom is of mild intensity, without interfering in the patient's activity
  2. The symptom is of moderate intensity, causing obvious discomfort to the patient
  3. The symptom is stated as very irritating and severe in intensity A Global Symptoms Score will be calculated by summing the intensities of all the three symptoms of vaginal atrophy in a certain time point, thus ranging between 0 and 9.
Time Frame: week 3 and week 12 vs baseline
Population: postmenopausal women
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 0.005% Estriol Vaginal Gel | Placebo Vaginal Gel
Number analyzed (Participants) | 50 | 11
score on a scale
  Change between baseline and week 3 | 3.0 [2.0 to 4.5] | 1.0 [0.5 to 3.0]
  Change between baseline and week 12 | 4.5 [3.0 to 7.0] | 2.0 [1.5 to 4.0]
Statistical Analysis 1: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Changes in total score of symptoms of vaginal atrophy from baseline to week 3; Test type: Other; p = 0.03, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Changes in total score of symptoms of vaginal atrophy from baseline to week 12; Test type: Other; p = 0.04, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Changes in Dryness of the Mucosa
Description: It will be scored by the investigator on a numerical scale in accordance with their presence and degree of severity as follows:
  0 Absence. The sign is not present.
  1. The sign is present and is considered a mild alteration
  2. The sign is present and is considered a moderate alteration
  3. The sign is present and is considered a severe alteration
Time Frame: week 3 and week 12 vs baseline
Population: postmenopausal women
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 0.005% Estriol Vaginal Gel | Placebo Vaginal Gel
Number analyzed (Participants) | 50 | 11
score on a scale
  Changes between baseline and week 3 | 2.0 [1.0 to 2.0] | 1.0 [0.0 to 1.0]
  Changes between baseline and week 12 | 2.0 [1.0 to 2.0] | 1.0 [0.0 to 1.0]
Statistical Analysis 1: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Changes in dryness of the mucosa between baseline and week 3; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Changes in dryness of the mucosa betweeen baseline and week 12; Test type: Other; p < 0.01, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Changes in Fragility of the Mucosa [Time Frame: Week 3 and Week 12 vs Baseline]
Description: as for outcome 12
Time Frame: from baseline to week 3 and 12
Population: Postmenopausal women
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 0.005% Estriol Vaginal Gel | Placebo Vaginal Gel
Number analyzed (Participants) | 50 | 11
score on a scale
  Changes from baseline to week 3 | 1.0 [0.0 to 2.0] | 0.0 [0.0 to 1.0]
  Changes from baseline to week 12 | 1.5 [1.0 to 2.0] | 0.5 [0.0 to 1.0]
Statistical Analysis 1: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Changes in dryness of the mucosa between baseline and week 3; Test type: Other; p = 0.13, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Changes in dryness of the mucosa between baseline and week 12; Test type: Other; p < 0.01, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Changes in Vaginal Mucosa With Flattening of Folds or Thinning
Description: as for outcome 12
Time Frame: week 3 and week 12 vs baseline
Population: postmenopausal women
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 0.005% Estriol Vaginal Gel | Placebo Vaginal Gel
Number analyzed (Participants) | 50 | 11
score on a scale
  Change between baseline and week 3 | 1.0 [1.0 to 2.0] | 0.0 [0.0 to 0.0]
  Change between baseline and week 12 | 1.0 [1.0 to 2.0] | 0.0 [0.0 to 1.0]
Statistical Analysis 1: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Change from baseline to week 3; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Change from baseline to week 12; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Changes in Total Score of Signs of Vaginal Atrophy Between Week 3 and Week 12 to Baseline
Description: The signs evaluated Will be the following: vaginal mucosa with flattening of folds or thinning, dryness of the mucosa and Fragility of the mucosa.
  It will be scored by the investigator on a numerical scale in accordance with their presence and degree of severity as follows:
  0 Absence. The sign is not present.
  1. The sign is present and is considered a mild alteration
  2. The sign is present and is considered a moderate alteration
  3. The sign is present and is considered a severe alteration A Total Signs Score will be calculated by summing the intensities of all the three signs of vaginal atrophy in a certain time point, thus ranging between 0 and 9.
Time Frame: week 3 and week 12 vs baseline
Population: postmenopausal women
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 0.005% Estriol Vaginal Gel | Placebo Vaginal Gel
Number analyzed (Participants) | 50 | 11
score on a scale
  Change between baseline and week 3 | 4.0 [2.0 to 5.0] | 1.0 [0.0 to 2.0]
  Change between baseline and week 12 | 5.0 [4.0 to 6.0] | 1.0 [1.0 to 3.0]
Statistical Analysis 1: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Change in total score of signs between week 3 and baseline; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Change in total score of signs between week 12 and baseline; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Changes in Vaginal Maturation Value
Description: Vaginal cytology sample to evaluate the vaginal Maturation Value. For the cytologic evaluation, the number of parabasal, intermediate and superficial cells will be calculated in duplicate on 100 consecutive cells of vaginal cytology. The average of the two percentages obtained for each cell type will be calculated, which will serve to determine the maturation value (MV) based on the following formula:
  0.2 x (% parabasal) + 0.6 x (% intermediate) + 1.0 x (% superficial).
Time Frame: week 3 and week 12 vs baseline
Population: postmenopausal women
Measure: Median (Inter-Quartile Range); unit: % of cells
Arm/Group | 0.005% Estriol Vaginal Gel | Placebo Vaginal Gel
Number analyzed (Participants) | 50 | 11
% of cells
  Change between baseline and week 3 | -62.0 [-70.04 to -37.8] | -0.6 [-11.6 to 2.0]
  Change between baseline and week 12 | -37.2 [-55.0 to -5.4] | -1.0 [-36.4 to 1.4]
Statistical Analysis 1: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Change in maturation value from baseline to week 3; Test type: Other; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 0.005% Estriol Vaginal Gel vs Placebo Vaginal Gel; Change in maturation value from baseline to week 12; Test type: Other; p = 0.006, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: From baseline to last visit (up to 16 weeks)
Description: AE: Any new untoward medical occurrence or worsening of a pre-existing medical condition in a patient or clinical investigation subject administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment.
Arm/Group | 0.005% Estriol Vaginal Gel | Placebo Vaginal Gel
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/50 | 0/11
Other Adverse Events (participants affected / at risk) | 3/50 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.005% Estriol Vaginal Gel (N=50) | Placebo Vaginal Gel (N=11)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — An unrelated Serious adverse event (lymphoma) was reported but before study treatment administration
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.005% Estriol Vaginal Gel (N=50) | Placebo Vaginal Gel (N=11)
Urinary tract infection (Infections and infestations) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2014-11-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT02413008/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT02413008/SAP_001.pdf